CLINICAL TRIAL: NCT03090425
Title: Inflammatory/Familial Dilated Cardiomyopathy: Is There a Link to Autoimmune Diseases? TP9a of the KNHI Associated to the DZHK
Brief Title: Inflammatory/Familial Dilated Cardiomyopathy: Is There a Link to Autoimmune Diseases? TP9a
Acronym: Ikarius
Status: Completed | Type: Observational
Sponsor: Philipps University Marburg (Other)
Collaborators: Deutsches Zentrum für Herz-Kreislauf-Forschung (DZHK) (Other); Competence Network Heart Failure (Other)
Responsible Party: Principal Investigator, Sabine Pankuweit, Prof. Dr., Philipps University Marburg
Other Study IDs: 01 GI 0205 KKS 1108
Record Dates: First submitted 2017-03-14; First posted 2017-03-24 (Actual); Last update posted 2019-03-25 (Actual); Status verified 2019-03

CONDITIONS: Non Ischemic Cardiomyopathy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
In a hitherto ill-defined proportion of patients with inflammatory/familial cardiomyopathy, the phenotype dilative cardiomyopathy (DCM) is assumed to be the endstage of a multifactorial etiopathogenetic pathophysiology. Precipitating factors include enhanced autoimmunity, predisposition for viral infections, environmental factors in addition to a specific 'genetic background' of the individual patient. It is unresolved, whether the susceptibility to immunologically mediated myocardial damage reflects the presence of genetic risk factors shared by other autoimmune diseases, or is cardio-specific with individual predisposing factors. Aims of the project are the search for a genetic link or oredisposition to autoimmune diseases in patients with familial / inflammatory DCM.

DETAILED DESCRIPTION:
Epidemiological investigations in patients with autoimmune diseases have shown that in addition to a specific genetic alteration secondary inducing factors are responsible for the onset of the disease, which may lead to different phenotypes of autoimmune diseases in a single family. The working hypothesis has been derived that inflammatory DCM is the endstage of an autoimmune cardiac disease that goes along with the activation of succeptibility genes, which are common to other autoimmune diseases.

Original aims of the project were:

* inclusion of patients with dilated cardiomyopathy (ejection fraction <45%, left ventricular enddiastolic diameter > 56mm) and in addition
* the inclusion of all relevant data regarding a possible familial, infectious or autoimmune etiology of the disease. A questionnaire was added to the CRFs, in order to ascertain data regarding a possible familial history for each patient not only for cardiac diseases, but also for autoimmune disorders. A pedigree of all patients was drawn. Data regarding a possible infectious or inflammatory etiology of the disease are available by investigation of the endomyocardial biopsy and peripheral blood. All data were included in the CRF. Derived from the data base, the biopsy and serum bank, further aims of the project are the search for a genetic link or genetic predisposition for autoimmune diseases in patients with DCM, especially inflammatory diseases.

To reach these aims, peripheral blood of all included patients was sent to the biomaterial bank in Berlin. DNA extracted from peripheral blood was investigated for the detection of genetic abnormalities in the genes for structural proteins, which are known to be associated with DCM. In addition, screening was done for several candidate genes in endomyocardial biopsies of patients with DCM using microchip technology and the investigation for polymorphisms in the HLA class II DQ locus in the patient cohort. Data if this Investigation were correlated with clinical outcome of the patients, who clinically were followed in total for 10 years. Right now the 10 year follow-up is ongoing.

ELIGIBILITY:
Inclusion Criteria:

Patients between 18 and 70 years of age were included if they had a left ventricular ejection fraction of 45% and a left ventricular end-diastolic diameter >56 mm estimated by echocardiography with no evidence of significant valve disease.

Exclusion Criteria:

Coronary artery disease (>50% diameter luminal stenosis in one or more epicardial vessels) was excluded in all patients by means of coronary angiography. Moreover, patients were excluded from the study if they demonstrated one or more of the following parameters: peripartum cardiomyopathy, history of myocardial infarction, severe systemic hypertension, alcohol abuse, and drug dependency.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with non ischemic DCM: All patients underwent a careful history and clinical examination aswell as laboratory studies and echocardiographic assessment with 2-dimensional echocardiography. The diagnosis of DCM was made according to criteria of the position statement from the European Society of Cardiology working group on myocardial and pericardial diseases
Sampling Method: Probability Sample
Enrollment: 320 (Actual)
Dates: Start 2016-06 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Genotype - phenotype correlation in patients with DCM of different etiology | 10-year clinical Follow-up will be performed from 12/2016 until June 2018
  Correlation of different clinical and genetic marker with outcome (ejection fraction, left ventricular Diameter, composite of all-cause mortality or heart Transplantation

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Karatolios K, Holzendorf V, Richter A, Schieffer B, Pankuweit S; Competence Network Heart Failure Germany. Long-term outcome and predictors of outcome in patients with non-ischemic dilated cardiomyopathy. Int J Cardiol. 2016 Oct 1;220:608-12. doi: 10.1016/j.ijcard.2016.06.167. Epub 2016 Jun 26. PMID 27390998
- [Background] Pankuweit S, Ruppert V, Jonsdottir T, Muller HH, Meyer T; German Competence Network of Heart Failure. The HLA class II allele DQB1 0309 is associated with dilated cardiomyopathy. Gene. 2013 Dec 1;531(2):180-3. doi: 10.1016/j.gene.2013.09.022. Epub 2013 Sep 16. PMID 24050898
- [Background] Meyer T, Ruppert V, Ackermann S, Richter A, Perrot A, Sperling SR, Posch MG, Maisch B, Pankuweit S; German Competence Network Heart Failure. Novel mutations in the sarcomeric protein myopalladin in patients with dilated cardiomyopathy. Eur J Hum Genet. 2013 Mar;21(3):294-300. doi: 10.1038/ejhg.2012.173. Epub 2012 Aug 15. PMID 22892539
- [Background] Waldmuller S, Erdmann J, Binner P, Gelbrich G, Pankuweit S, Geier C, Timmermann B, Haremza J, Perrot A, Scheer S, Wachter R, Schulze-Waltrup N, Dermintzoglou A, Schonberger J, Zeh W, Jurmann B, Brodherr T, Borgel J, Farr M, Milting H, Blankenfeldt W, Reinhardt R, Ozcelik C, Osterziel KJ, Loeffler M, Maisch B, Regitz-Zagrosek V, Schunkert H, Scheffold T; German Competence Network Heart Failure. Novel correlations between the genotype and the phenotype of hypertrophic and dilated cardiomyopathy: results from the German Competence Network Heart Failure. Eur J Heart Fail. 2011 Nov;13(11):1185-92. doi: 10.1093/eurjhf/hfr074. Epub 2011 Jul 12. PMID 21750094
- [Background] Ruppert V, Meyer T, Struwe C, Petersen J, Perrot A, Posch MG, Ozcelik C, Richter A, Maisch B, Pankuweit S; German Heart Failure Network. Evidence for CTLA4 as a susceptibility gene for dilated cardiomyopathy. Eur J Hum Genet. 2010 Jun;18(6):694-9. doi: 10.1038/ejhg.2010.3. Epub 2010 Feb 10. PMID 20145677
- [Result] Pankuweit S, Luers C, Richter A, Ruppert V, Gelbrich G, Maisch B; German Competence Network Heart Failure. Influence of different aetiologies on clinical course and outcome in patients with dilated cardiomyopathy. Eur J Clin Invest. 2015 Sep;45(9):906-17. doi: 10.1111/eci.12483. Epub 2015 Aug 6. PMID 26094644
- [Derived] Binas D, Daniel H, Richter A, Ruppert V, Schluter KD, Schieffer B, Pankuweit S. The prognostic value of sST2 and galectin-3 considering different aetiologies in non-ischaemic heart failure. Open Heart. 2018 Feb 26;5(1):e000750. doi: 10.1136/openhrt-2017-000750. eCollection 2018. PMID 29531765